CLINICAL TRIAL: NCT06657482
Title: Effects of Delayed School Start Times on Sleep, Mental Health, and Academic Performance Among Norwegian Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REK Vest 606094
Record Dates: First submitted 2024-07-03; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Sleep; Sleep Disorders, Circadian Rhythm; Psychiatric Disorder; Sleepiness, Daytime
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Mental Disorders; Disorders of Excessive Somnolence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed school start times on Mondays and Tuesdays (intervention condition) (Experimental): Two hour delay in school start time on Mondays and one hour delay on Tuesdays. Ordinary school start time (8:15 ± 15 min) for the rest of the week.
  Interventions: Behavioral: Delayed school start time
- Ordinary school start time all weekdays (control condition) (No Intervention): Ordinary school start time (8:15 ± 15 min) all school days

INTERVENTIONS:
Behavioral: Delayed school start time — The intervention group will start school two hours later on Mondays (at 10.15 ± 15 min) and one hour later on Tuesdays (9.15 ± 15 min) and to ordinary school start time (8.15 ± 15 min) for the rest of the week
  Arms: Delayed school start times on Mondays and Tuesdays (intervention condition)

SUMMARY:
The aim is to investigate whether later school start times have positive effects on high school students' sleep patterns, mental health and daytime functioning.

DETAILED DESCRIPTION:
The current study is a randomized controlled study investigating whether later school start times on Mondays and Tuesdays have positive impact on high school students' sleep patterns, mental health, and daytime functioning. 1st year high school students are randomly assigned to classes starting either two hours later on Mondays and one hour later on Tuesday and ordinary school start times (8:15 ± 15 min) for the rest of the week, or to classes starting at regularly school start times (8:15 ± 15 min.) all weekdays. The students will be invited to respond to a web-based survey assessing sleep, mental health, and daytime functioning by the beginning and end of the school year. Official school grades and school absence data will be collected through the county administration for consenting students. Cognitive tests and objective sleep record through Somnofy are planned for a subgroup by the end of the 2024-25 school year. The study will last for two school years and involve two different cohorts of 1st year high school students.

ELIGIBILITY:
Inclusion Criteria:

* 1st year high school students at study preparatory program of participating schools

Exclusion Criteria:

* Parent consent not obtained/documented for participants under 16 years

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Average sleep duration on school days | Baseline and at the end of the school year (at about 8 months follow-up)
  Average sleep duration across the arms will be calculated using the Munich ChronoType Questionnaire (MCTQ), adjusted for nocturnal awakenings
Preferred school start time (late vs. early Mondays and Tuesdays) | At the end of the school year (at about 8 months follow-up)
  A conditioned item asking how satisfied the students are starting early or later on Mondays and Tuesdays, or ranging from "Very satisfied" to "very dissatisfied", will be included.
Daytime sleepiness on school days | CADSS: Baseline and at the end of the school year (at about 8 months follow-up). KSS: At the end of the school year (at about 8 months follow-up)-up
  Daytime sleepiness will be assessed based on the Karolinska Sleepiness Scale (KSS; adjusted to target sleepiness on each weekday) and The Chinese adolescent daytime sleepiness scale (CADSS).

SECONDARY OUTCOMES:
School absence and academic performance (self-reported and objective) | Self-reported data: Baseline and end of school year. Objective data: At the end of the school year (at about 8 months follow-up)-up
  Data gathered from school authorities.
Mental health | Baseline and at the end of the school year (at about 8 months follow-up)
  Anxiety and depression will be assessed during the past two weeks using the Generalized Anxiety Disorder-7 and the Patient Health Questionnaire-9, respectively.
Social jetlag | Baseline and at the end of the school year (at about 8 months follow-up)
  Social jetlag, calculated as the discrepancy in sleep timing on free vs. weekdays, will be calculated based on the MCTQ
Sleep duration, school days with early vs. late start | At the end of the school year (at about 8 months follow-up)
  Sleep duration for late starting days will be compared with early starting days

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Bjorvatn, Principal Investigator — Department of Global Public Health and Primary Care, University of Bergen, Norway
Locations (1):
- University of Bergen, Bergen, Vestland, Norway